CLINICAL TRIAL: NCT03899779
Title: Face-to-face Versus Online Hypnotherapy for the Treatment of Irritable Bowel Syndrome, According to a Non-inferiority Design. Three-armed Randomized Controlled Trial.
Brief Title: Face-to-face Versus Online Hypnotherapy for the Treatment of Irritable Bowel Syndrome
Acronym: FORTITUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL67607.068.18; 852001924 (Other Grant/Funding Number: ZonMw); METC18-037 (Other: METC azM/UM)
Record Dates: First submitted 2019-02-13; First posted 2019-04-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Face-to-face hypnotherapy (Active Comparator): 12 weeks treatment with face-to-face hypnotherapy (6 individual, bi-weekly sessions)
  Interventions: Other: Face-to-face hypnotherapy
- Online hypnotherapy (Experimental): 12 weeks treatment with online hypnotherapy
  Interventions: Other: Online hypnotherapy
- Online psychoeducation (Active Comparator): 12 weeks treatment with online psychoeducation
  Interventions: Other: Online psychoeducation

INTERVENTIONS:
Other: Face-to-face hypnotherapy — 12 weeks treatment with face-to-face hypnotherapy (6 individual, bi-weekly sessions)
  Arms: Face-to-face hypnotherapy
Other: Online hypnotherapy — 12 weeks treatment with online hypnotherapy
  Arms: Online hypnotherapy
Other: Online psychoeducation — 12 weeks treatment with online psychoeducation
  Arms: Online psychoeducation

SUMMARY:
Psychological therapies are effective in reducing irritable bowel syndrome (IBS) symptom severity and increasing quality of life and are recommended for the management of IBS by guidelines. Evidence appears strongest for the efficacy of hypnotherapy as psychological treatment. However, therapist-led interventions are time consuming and relatively costly. Approaches based on e-health are cost saving and appear more attractive to patients as no visits to a therapist are necessary. Therefore, the investigators plan to conduct a multicentre randomised controlled trial to examine whether the effectiveness of online hypnotherapy is non-inferior compared to individual face-to-face hypnotherapy delivered by a therapist, according to current FDA guidelines. Online psychoeducation will be used as control condition. In addition, the investigators hypothesize that treatment with online hypnotherapy is a more cost-effective therapy than face-to-face hypnotherapy in IBS patients.

ELIGIBILITY:
Inclusion criteria:

* Age 16-75 years
* A diagnosis of IBS according to the Rome IV criteria
* In the presence of alarm symptoms, such as rectal blood loss, weight loss, anemia, first onset of symptoms above 50 years of age, patients will be first referred for further investigation by their treating physician to exclude organic disorders, conform current Dutch guidelines for IBS.
* Women in fertile age must use contraception or be postmenopausal for at least two years.

Exclusion criteria:

* Insufficient command of the Dutch language
* No access to internet
* Evidence of current anxiety and/or depression disorder as defined by a score ≥10 on the GAD-7 and/or PHQ-9 questionnaire. In this case it is conceivable that the IBS symptoms are strongly related to psychopathology for which different treatment might be more appropriate.
* History of ulcerative colitis, Crohn's disease, coeliac disease or significant liver disease
* Major surgery to the lower gastrointestinal tract, such as partial or total colectomy, small bowel resection or partial or total gastrectomy
* Past or present radiotherapy to the abdomen
* Current pregnancy or lactation
* Using of psychoactive medication in case there's no stable dose for at least 3 months prior to inclusion
* Use of over-the-counter or prescription antidiarrheals, analgesics and laxatives (only be allowed as specific rescue medication)
* Hypnotherapy treatment received in the last 3 months prior to inclusion
* Using more than 20 units of alcohol per week
* Using drugs of abuse

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-06-29 (Actual)

PRIMARY OUTCOMES:
Abdominal pain response rate after 12 weeks of treatment | 12 weeks
  A responder is defined as a patient who experiences at least a 30 percent decrease in the weekly average of worst daily abdominal pain (measured daily, on an 11 point NRS) compared to baseline weekly average in at least 50 percent of the weeks in which the treatment in given.

SECONDARY OUTCOMES:
Degree of relief response rate after 12 weeks of treatment | 12 weeks
  A responder is defined as a patient who experiences a weekly relief of 1 or 2 (on a 7 point NRS) in at least 50 percent of the weeks in which treatment is given.
Improvement of symptom severity | 16 weeks
  determined by the Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) by 50 points or more [IBS-SSS, minimum score 0, maximum score 500]
Indirect costs | 16 weeks and after 6 months and 1 year follow-up
  determined by Productivity Cost Questionnaire (PCQ) (savings from increased work productivity)
Direct costs | 16 weeks and after 6 months and 1 year follow-up
  determined by Medical Consumption Questionnaire (MCQ) (savings from reduced medical resource use)
General Quality of life (by EQ-5D) | 16 weeks and after 6 months and 1 year follow-up
  Determined by the Euro-Quality of Life - 5 domains (EQ-5D-5L) (change from baseline)
IBS related Quality of life (by IBS-QoL) | 16 weeks and after 6 months and 1 year follow-up
  Determined by IBS Quality of Life (IBS-QoL) (change from baseline) [IBS-QoL, minimum score: 0, maximum score 100]
Use of over the counter medication and rescue medication | 12 and 16 weeks
  As reported via digital diary (mobile phone application)
Number and severity of side effects | 12 and 16 weeks
  As reported via digital diary (mobile phone application)
Expectation | 16 weeks
  Response rates in relation to patient expectation prior to the start of treatment
Response rates in relation to comorbid anxiety | 16 weeks and after 6 months and 1 year follow-up
  Assessed with the use of the Generalized Anxiety Disorder-7 (GAD-7). [GAD-7 minimum score: 0, maximum score: 21]
Response rates in relation to comorbid depression | 16 weeks and after 6 months and 1 year follow-up
  Assessed with the use of the Patient Health Questionnaire-9 (PHQ-9). [PHQ-9 minimum score: 0, maximum score: 21]

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keszthelyi, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (6):
- Netherlands (6):
  - Gelderse Vallei, Ede, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Bernhoven, Uden, North Brabant
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Martini Ziekenhuis, Groningen, Provincie Groningen